CLINICAL TRIAL: NCT00496860
Title: Phase I Study of ALT-801 in Patients With Progressive Metastatic Malignancies
Brief Title: Safety and Efficacy Study of ALT-801 to Treat Progressive Metastatic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-01-06
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Progressive Metastatic Malignancies
Keywords: cancer; p53; immunotherapy; targeted; metastatic; malignancy; malignancies; interleukin-2; IL-2; fusion protein; antitumor; melanoma; renal cancer; lung cancer; kidney cancer; breast cancer; colorectal cancer; colon cancer; renal cell carcinoma; advanced cancer; head and neck cancer; breast tumors; cancer of head and neck; esophagus cancer; lymphoma; ovarian cancer; ovary cancer; bladder cancer; stomach cancer; TCR; T-cell receptor; P53 gene; p53 tumor suppressor protein
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Melanoma; Kidney Neoplasms; Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Head and Neck Neoplasms; Esophageal Neoplasms; Lymphoma; Ovarian Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms | interventions — ALT-801

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ALT-801 — Dose escalation (0.015 mg/kg, 0.04 mg/kg, 0.08 mg/kg, 0.12 mg/kg, 0.14 mg/kg, 0.16 mg/kg), intravenous infusions, two treatment cycle, each cycle with 4 daily on-dose infusion, 10 days rest between cycles.

SUMMARY:
This is a Phase 1, open-labeled, non-randomized, multi-center, competitive enrollment and dose-escalation study of ALT-801, the study drug. The purpose of this study is to evaluate the safety, determine the maximum-tolerated dose (MTD) and characterize the pharmacokinetic profile of ALT-801 in previously treated patients with progressive metastatic malignancies. ALT-801, a recombinant fusion protein with a interleukin-2 (IL-2) component, has a targeting mechanism that recognizes tumor cells with a specific tumor marker.

DETAILED DESCRIPTION:
Most current cancer treatment strategies involve the use of chemotherapeutic or biological drugs that exhibit variable efficacy and considerable toxicity. The limitations are often the result of the adverse side effects of the therapeutic drug on normal tissues. One approach to control these effects is to target the therapy to the tumor site. Of the identified tumor antigens, the human p53 tumor suppressor protein is overexpressed in a wide range of human malignancies. p53 is an intracellular tumor suppressor protein that acts to arrest the proliferation of cells. When mutated, it loses its ability to suppress abnormal proliferation and exhibits a longer half-life than the wild-type protein, allowing for its accumulation in tumors. In addition, p53 overexpression correlates with tumor transformation and aggression and is associated with lower overall survival rates and resistance to chemotherapeutic intervention in cancer patients. Therefore, p53 appears to be a marker for a considerable number of human malignancies and represents a good target for immunotherapeutics. However, p53 cannot be used as a target for antibodies because it is not displayed independently on the cell surface. Instead, the p53 protein is processed intracellularly into peptide fragments that are then displayed on the cell surface in the context of major histocompatibility complex (MHC). These peptide/MHC complexes are recognized by T-cells via their T-cell receptors (TCRs). Recently it has been confirmed that the peptide fragment is significantly elevated in a wide range of human tumor tissues, particularly in melanoma, renal, lung, breast, colorectal, bladder, ovary, stomach, esophagus, lymphoma, liver, leukemia, and head & neck cancer. Targeted approaches to concentrate therapeutic cytokines at the tumor sites that express p53 could provide considerable advantages over current treatment.

Interleukin-2 (IL-2) is a well-characterized growth factor for immune effector cells which play critical roles in tumor control and rejection. A recombinant human IL-2 has been approved for treating metastatic melanoma and renal cell carcinoma. However, the major drawback of IL-2 therapy is its severe systemic toxicity. As a result, use of high dose IL-2 is limited to specialized programs with experienced personnel and it is generally offered to patients who are responsive and have excellent organ function. Thus, there is a critical need for innovative strategies that enhance the effects of IL-2 or reduce its toxicity without compromising clinical benefits.

The study drug, ALT-801, is a biologic compound composed of interleukin-2 (IL-2) genetically fused to a humanized soluble T-cell receptor directed against the p53-derived antigen. This study is to evaluate whether directing IL-2 activity using ALT-801 to the patient's tumor sites that overexpress p53 results in clinical benefits.

The study drug will be administered by bolus intravenous infusion in an in-patient hospital setting under the supervision of a qualified physician experienced in the use of anti-cancer agents including high dose IL-2. An intensive care facility and specialists skilled in cardiopulmonary or intensive care medicine must be available. There are two treatment cycles. For each treatment cycle, patients will be admitted to the hospital, remain in the hospital during the study drug infusion period, and be discharged from the hospital the day after the last infusion at the Principal Investigator's discretion. There is a 10-day resting period between the treatment cycles. Tumor assessments will be done at weeks 7 and 11 after starting the study drug.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARACTERISTICS:

* Locally advanced or metastatic malignancies
* Histologically or cytologically confirmed
* Evaluable
* Surgically and medically incurable
* Not responding to standard therapy or no other standard therapy exists
* Human leukocyte antigen (HLA)-A2.1/p53 positive

PRIOR/CONCURRENT THERAPY:

* No prior Proleukin therapy within one year
* No concurrent radiotherapy, chemotherapy, or other immunotherapy
* More than 4 weeks since prior major radiotherapy
* More than 4 weeks since prior cytotoxic therapy
* More than 6 weeks since prior nitrosoureas therapy
* More than 8 weeks since prior monoclonal antibody therapy

PATIENT CHARACTERISTICS:

Life expectancy

* > 3 months

Performance status

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1

Bone marrow reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1,500/microliters (uL)
* Platelets ≥100,000/uL
* Hemoglobin ≥ 10g/dL

Renal function

* Serum creatinine ≤ 1.5 X Upper limit of normal (ULN)

Hepatic function

* Total bilirubin ≤ 1.5 X ULN
* Aspartate Aminotransferase (AST) ≤ 2.5 X ULN
* Alkaline phosphatase ≤ 2.5 X ULN
* Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 X ULN
* Activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN

Cardiovascular

* May be safely tapered off anti-hypertensives if currently on anti-hypertensives
* New York Heart Association classification I or II
* No congestive heart failure <6 months
* No unstable angina pectoris <6 months
* No myocardial infarction <6 months
* No history of ventricular arrhythmias
* Normal cardiac stress test required if any of the following is present:

  * Over age 50
  * History of abnormal EKG
  * Symptoms of cardiac ischemia or arrhythmia

Pulmonary

* Normal pulmonary function test (FEV1 ≥ 75% of predicted value) if any of the following is present:

  * Prolonged history of cigarette smoking
  * Symptoms of respiratory dysfunction

Other

* No known autoimmune disease
* No known HIV positive
* No psychiatric illness/social situations that would limit study compliance
* No history or evidence of central nervous system (CNS) disease
* No active systemic infection requiring parental antibiotic therapy
* No systemic steroid therapy required
* No prior organ allograft
* Not receiving other investigational agents
* Not receiving chronic medication for asthma
* Not pregnant or nursing
* Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado, Anschutz Cancer Pavillion, Aurora, Colorado
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Washington, Seattle Cancer Care Center, Seattle, Washington

REFERENCES:
- [Derived] Fishman MN, Thompson JA, Pennock GK, Gonzalez R, Diez LM, Daud AI, Weber JS, Huang BY, Tang S, Rhode PR, Wong HC. Phase I trial of ALT-801, an interleukin-2/T-cell receptor fusion protein targeting p53 (aa264-272)/HLA-A*0201 complex, in patients with advanced malignancies. Clin Cancer Res. 2011 Dec 15;17(24):7765-75. doi: 10.1158/1078-0432.CCR-11-1817. Epub 2011 Oct 12. PMID 21994418
- See also: Altor Bioscience Corporation, Miramar, Florida, US — http://www.altorbioscience.com
- See also: H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, US — http://www.moffitt.org
- See also: MD Anderson Cancer Center Orlando — http://www.orlandoregional.org/mdanderson/index.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 08-2007 and 05-2009, 118 patients were consented and screened, 56 were Human leukocyte antigen (HLA)-A2 positive and had tumor specimens that were positive for target p53 (aa 264-272)/HLA-A*0201 complex. Thirty HLA-A2-positive patients with p53/HLA-A*0201 tumors either withdrew consent or did not meet other inclusion/exclusion criteria.
Groups:
- ALT-801 0.015 mg/kg/Dose: 0.015 mg/kg/dose of ALT-801
- ALT-801 0.040 mg/kg/ Dose: 0.040 mg/kg/dose of ALT-801
- ALT-801 0.080 mg/kg/Dose: 0.080 mg/kg/dose of ALT-801
Period: Overall Study
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/ Dose | ALT-801 0.080 mg/kg/Dose
Started | 4 | 16 | 6
Completed | 3 | 15 | 6
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ALT-801 0.040 mg/kg/Dose: 0.040 mg/kg/dose of ALT-801
- Total: Total of all reporting groups
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose | Total
Number analyzed (Participants) | 4 | 16 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 15 | 5 | 22
  >=65 years | 2 | 1 | 1 | 4
Age Continuous [Median (Full Range); unit: years] | 65 [50 to 79] | 51 [27 to 72] | 58 [53 to 65] | 54 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 1 | 9
  Male | 2 | 10 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 15 | 6 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Toxicity of ALT-801 in Patients With Progressive Metastatic Malignancies
Description: Number of serious adverse events per cohort
Time Frame: 18 months
Measure: Number; unit: Events
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Number analyzed (Participants) | 4 | 16 | 6
Events | 0 | 2 | 4

2. Primary Outcome: The Maximum-tolerated Dose (MTD) of ALT-801
Description: Number of dose limiting toxicities (DLTs). A DLT is a toxicity that results in patient withdrawal from the study as defined in the protocol.
Time Frame: 18 months
Measure: Number; unit: events
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Number analyzed (Participants) | 4 | 16 | 6
events | 0 | 1 | 2

3. Secondary Outcome: Clinical Antitumor Response to ALT-801
Description: Number of subjects with a complete response (CR), partial response (PR) or stable disease (SD). CR is defined as disappearance of all tumor lesions selected for measurement. PR is defined as at least 30% decrease in the sum of all tumor lesions selected for measurement. Stable disease is defined as neither sufficient tumor shrinkage to qualify for PR nor sufficient tumor increase to qualify for progressive disease (PD) which is defined as at least 20% increase the sum of the all tumor lesions selected for measurement.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Number analyzed (Participants) | 4 | 16 | 6
participants | 2 | 5 | 3

4. Secondary Outcome: ALT-801 Induced Cell-mediated Immune Responses
Description: Number of tumor-responsive (interferon-gamma positive (IFNg+)) immune cells in blood post dosing
Time Frame: 24 months
Measure: Mean (Standard Error); unit: IFNg spots per million PMBCs
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Number analyzed (Participants) | 3 | 16 | 6
IFNg spots per million PMBCs | 6433 (2847) | 9117 (1671) | 1125 (163)

5. Secondary Outcome: Immunogenicity of ALT-801
Description: Titer of anti-drug Abs at week 4
Time Frame: 24 months
Measure: Mean (Standard Error); unit: titer
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Number analyzed (Participants) | 3 | 16 | 6
titer | 347 (103) | 5483 (2310) | 762 (97)

ADVERSE EVENTS:
Arm/Group | ALT-801 0.015 mg/kg/Dose | ALT-801 0.040 mg/kg/Dose | ALT-801 0.080 mg/kg/Dose
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/16 | 4/6
Other Adverse Events (participants affected / at risk) | 4/4 | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALT-801 0.015 mg/kg/Dose (N=4) | ALT-801 0.040 mg/kg/Dose (N=16) | ALT-801 0.080 mg/kg/Dose (N=6)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death-NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALT-801 0.015 mg/kg/Dose (N=4) | ALT-801 0.040 mg/kg/Dose (N=16) | ALT-801 0.080 mg/kg/Dose (N=6)
Rhinitis (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 12 (12) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 3 (3) | 10 (10) | 4 (4)
Supraventricular arrhythmia - Sinus tachycardia (Cardiac disorders) | 0 (0) | 8 (8) | 3 (3)
Ventricular arrhythmia - Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 9 (9) | 5 (5)
INR (Investigations) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 9 (9) | 0 (0)
Fever (General disorders) | 4 (4) | 16 (16) | 6 (6)
Insomnia (General disorders) | 0 (0) | 6 (6) | 0 (0)
Rigors/chills (General disorders) | 2 (2) | 14 (14) | 6 (6)
Weight gain (General disorders) | 2 (2) | 2 (2) | 2 (2)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 2 (2)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 10 (10) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (10) | 1 (1)
Infection with normal ANC (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Edema: trunk/genital (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1) | 6 (6) | 3 (3)
ALT (Investigations) | 1 (1) | 2 (2) | 0 (0)
AST (Investigations) | 1 (1) | 5 (5) | 0 (0)
Bicarbonate, serum-low (Investigations) | 0 (0) | 1 (1) | 1 (1)
Bilirubin (Investigations) | 1 (1) | 4 (4) | 2 (2)
Creatinine (Investigations) | 0 (0) | 3 (3) | 3 (3)
Hyperglycemia (Investigations) | 0 (0) | 5 (5) | 1 (1)
Hyperkalemia (Investigations) | 0 (0) | 2 (2) | 1 (1)
Hypermagnesemia (Investigations) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminemia (Investigations) | 3 (3) | 16 (16) | 6 (6)
Hypocalcemia (Investigations) | 3 (3) | 12 (12) | 5 (5)
Hypokalemia (Investigations) | 2 (2) | 8 (8) | 1 (1)
Hypomagnesemia (Investigations) | 1 (1) | 6 (6) | 4 (4)
Hyponatremia (Investigations) | 2 (2) | 13 (13) | 4 (4)
Hypophosphatemia (Investigations) | 2 (2) | 15 (15) | 4 (4)
Proteinuria (Investigations) | 0 (0) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6) | 0 (0)
Mood alteration (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Pain - Musculoskeletal (General disorders) | 1 (1) | 4 (4) | 3 (3)
Pain - Neurology (General disorders) | 0 (0) | 7 (7) | 0 (0)
Pain - Other (General disorders) | 0 (0) | 2 (2) | 1 (1)
Pain - Pulmonary (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Renal - Other - Decreased urine output (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less